CLINICAL TRIAL: NCT04507347
Title: Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicentre Study to Evaluate the Efficacy and Safety of TRC041266 Compared to Placebo in Patients With Chronic Stable Heart Failure, an LVEF ≥40%, Moderate to Severe Diastolic Dysfunction and Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of TRC041266 in Patients With Heart Failure, LVEF ≥40%, Diastolic Dysfunction and Type 2 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant hence study withdrawn
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT/P004/HF/19/03_01
Record Dates: First submitted 2020-07-16; First posted 2020-08-11 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2020-08

CONDITIONS: Chronic Stable Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, Placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product (Experimental): Eligible participants will be randomized to receive test product, TRC041266 1500 mg twice daily for 48 weeks.
  Interventions: Drug: TRC041266
- Placebo product (Placebo Comparator): Eligible participants will be randomized to receive matching placebo twice daily for 48 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRC041266 — TRC041266 sachet 1500 mg strengths
  Arms: Test product
Drug: Placebo — TRC041266 sachet 1500 mg matching placebo
  Arms: Placebo product

SUMMARY:
This study will be conducted as a randomized, multi-centre, double-blind, parallel-group, placebo-controlled study in patients receiving SoC therapy. Eligible participants will be randomized in a ratio of 1:1 to receive either test product, TRC041266 1500 mg or matching placebo twice daily for 48 weeks

DETAILED DESCRIPTION:
HFpEF is associated with high morbidity and mortality and the prevalence is on the rise globally. Diabetics are at increased risk of developing HFpEF.

There is no evidence based therapy to improve the disease condition and its associated functional incapacity. Some of the recently concluded trials, PARAGON-HF, EMPERIAL-PRESERVED, failed to demonstrate benefit and it is regarded as an area with high unmet need.

Phase 2 results have demonstrated that in diabetic patients with heart failure having LVEF >30% and receiving guideline-indicated therapy with RAS inhibitors and β-blockers, TRC4186 has the potential to improve worsening of heart failure, functional status, cardiac diastolic function and has no adverse effect on cardiac mortality.

Therefore, TRC041266, the decanoic acid co-crystal of TRC4186 is an innovative product for the management of heart failure with LVEF≥40% in diabetic patients which is expected to modify the underlying disease at multiple levels and confer benefit as add-on to standard of care.

The current phase 3 study has been planned based on the results of the phase 2 trial which demonstrated that the TRC4186 2000 mg/day (in two divided doses; BD) administered orally for 48 weeks resulted in significant improvement in QoL measured by PD-MLHFQ, diastolic dysfunction measured by E/e' and reduction in HF hospitalization.

The dose level to be used in the present study is based on the assessment of safety, efficacy and PK data obtained from phase 1 and 2 studies. In the phase 2 study, a dose response was observed with a trend towards improvement at 500 mg/day dose of TRC4186, and clinically and statistically significant improvement was seen at 2000 mg/day (1000 mg BD). There was plateauing of the response beyond the dose of 2000 mg/day. Hence, the choice of optimal dose of TRC4186 being considered is lower than 2000 mg/day and in between 500 and 2000 mg/day, i.e., 1500 mg/day (750 mg BD). The total daily dose of TRC041266 which would be equivalent to 1500 mg/day of TRC4186, is TRC041266 3000 mg/day, to be administered in two divided doses,i.e., 1500 mg BD.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 40-70 years (both inclusive)
2. Type 2 diabetes mellitus on stable hypoglycemic therapy for >1 month
3. Diagnosed with heart failure* according to 2016 ESC Guidelines for Chronic Heart Failure for at least 6 months and receiving SoC for at least 3 months

   *HF - a clinical syndrome characterized by typical symptoms (e.g. breathlessness, ankle swelling and fatigue) that may be accompanied by signs (e.g. elevated jugular venous pressure, pulmonary crackles and peripheral edema) caused by a structural and/or functional cardiac abnormality, resulting in a reduced cardiac output and/or elevated intra-cardiac pressures at rest or during stress
4. Participants with LVEF ≥40% including HFpEF according to ESC criteria, diagnosed by ECHO, confirmed by core ECHO laboratory AND having moderate to severe diastolic dysfunction as described in 'Classification of Diastolic Dysfunction'
5. NT-proBNP (N-terminal fragment of brain natriuretic peptide) 250-3500 pg/mL (both inclusive) For participants who have atrial fibrillation, the inclusion qualification would be 750- 3500 pg/ml (both inclusive)
6. Treatment with stable# doses of loop diuretics for >1 month at a daily dose of furosemide of ≥40 mg or equivalent (1 mg of bumetanide or 10 mg of torasemide) or alternatively, 20 mg furosemide + mineralocorticoid receptor antagonist or equivalent (0.5 mg of bumetanide + mineralocorticoid receptor antagonist or 5 mg of torasemide + mineralocorticoid receptor antagonist) or equivalent as per the regional SoC
7. On stable# doses of beta-blockers for >1 month

   * No exceptions are allowed to the above rule if LVEF is ≤50% OR the patient has coronary artery disease,
   * If LVEF is >50% and the patient is NOT KNOWN to have coronary disease, they may be included if they are not taking beta-blockers provided there is no indication to use them such as rate control for atrial fibrillation or hypertension
8. Participants willing to give written informed consent (prior to any study-related procedures being performed) and able to adhere to the study restrictions and assessments schedule

   * stable = a dose no lower than half the current dose and not greater than double the current dose

Exclusion Criteria:

1. Known hypersensitivity to any ingredient of the study medication
2. Heart failure caused by myocarditis, cor-pulmonale, congenital heart disease,constrictive pericarditis, idiopathic hypertrophic or restrictive cardiomyopathy, amyloid heart disease or rheumatic heart disease
3. Significant valvular heart disease including severe mitral regurgitation or left ventricular (LV) aneurysm as judged by the investigator and/or echo core-laboratory
4. History of MI, CABG surgery, PCI or other major surgery, stroke or TIA in past 6 months
5. Patients who are anticipated to require coronary revascularization; patients with angina must be evaluated by a cardiologist to determine the need for revascularization
6. NYHA class IV
7. A score of less than 12 points on adequately explained and administered MLHFQ points 2, 3, 4, 5, 7, 8, 12 and 13
8. Hospitalization for heart failure with overnight stay in the past 3 months
9. Participants with symptomatic or sustained VT* in the past 6 months and planned for cardiac resynchronization therapy (CRT) or implantation of ICD for the duration of the study.

   * Participant with symptomatic or sustained VT having an implantable cardioverter defibrillator (ICD) can be included in the study.
10. Atrial fibrillation or flutter with a resting ventricular rate >110 beats per minute
11. Unable to walk or has any contraindication to 6-minute walk test or those in whom longest distance walked in supervised 6 minutes (6MWTD) at baseline was <100 m or >350m
12. Systolic BP < 100 mmHg or ≥ 160 mmHg or Diastolic BP ≥ 100 mmHg at screening
13. Hb <12 g/dL
14. HbA1c >11%
15. eGFR <30 mL/min/1.73m2 (calculated by Modification of Diet in Renal Disease formula) [eGFR (mL/min/1.73 m²) = 175 × (Scr)-1.154 × (Age)-0.203 × (0.742 if female) × (1.212 if African American) (conventional units)]
16. Liver enzymes (AST or ALT) exceeding 3 times the upper limit of normal range at screening and considered clinically significant by the investigator
17. Current hyponatremia (Na+ <130 mmol/L) or hyperkalemia (K+ >5.5 mmol/L)
18. Participants on insulin as monotherapy for diabetes
19. History of gastrointestinal disorder (e.g. malabsorption syndrome) that could interfere with study drug absorption
20. Known to have positive test for HIV, Hepatitis B, Hepatitis C at the time of screening
21. History of malignancy in last 3 years other than basal cell carcinoma
22. Pregnant or lactating women, or female of childbearing potential, who are neither surgically sterilized nor willing to use reliable contraceptive methods (double barrier methods or intrauterine device)
23. Men with partners of childbearing potential not willing to use reliable contraception methods
24. Current participation (including prior 30 days) in any other therapeutic clinical trial
25. In the opinion of the investigator, any finding which would interfere with the objectives of the study, patient is unable to cooperate with any study procedures, unlikely to adhere to the study procedures, keep appointments, or plan to relocate during the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Primary composite endpoint consisting of incidence of cardiac mortality and/or number of worsening of heart failure and/or change from baseline to week 48 in functional capacity | 48 weeks
  Worsening of heart failure will be comprising of hospitalization for heart failure, or emergency visits for heart failure, or sustained increase in dose of diuretics
  Functional capacity shall be assessed by Physical Dimension-Minnesota Living with Heart Failure Questionnaire, and supervised 6-minute walk distance (measured in meters)

IPD SHARING:
Plan to Share IPD: No